CLINICAL TRIAL: NCT05316558
Title: Body Confident Coaching: Acceptability Testing of a Web-Based Body Image Intervention for Coaches of Adolescent Girls
Brief Title: Web-Based Body Image Intervention for Coaches of Adolescent Girls - Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the West of England (Other)
Collaborators: Unilever R&D (Industry); Nike (Industry); Laureus (Unknown); Tucker Center for Research on Girls & Women in Sport (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HAS.21.03.120b
Record Dates: First submitted 2022-03-18; First posted 2022-04-07 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Intervention; Waitlist Control
Keywords: Body image; Athletes; Girls; Coaches; Web-based; Coach education

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Body Confident Coaching (Experimental): Participants in the intervention condition will take part in an online program consisting of five modules over two weeks.
  Interventions: Behavioral: Body Confident Coaching
- Waitlist control (No Intervention): Participants will not be explicitly told their study condition, although they will be made aware of the assessment time points and whether they receive the intervention between T1 and T2 (intervention) or after T2 (waitlist control). Following completion of post-intervention assessments (T2), the control condition will participate in the intervention; but, they will not be monitored or assessed.

INTERVENTIONS:
Behavioral: Body Confident Coaching — The Body Confident Coaching program is a five-module online program aimed at upskilling coaches in identifying and tackling body image concerns among girls in sport. Each module will take approximately 20 minutes to complete and consists of educational content, interactive elements (quizzes, checklists, opinion polls, reflective exercises), and additional resources.
  Arms: Body Confident Coaching

SUMMARY:
According to the World Health Organization, only 15% of 11-17-year-old girls meet the recommended daily physical movement guidelines (e.g., 60-minutes per day). Despite extensive research highlighting the protective factors associated with sport on both mental and physical health, body image concerns are a key barrier to girls' participation in and enjoyment of sport. Sports-related environments and society more broadly further exacerbate these concerns through harmful gender stereotypes that perpetuate female objectification, discrimination, and harassment. This includes the promotion of unrealistic and sexualized appearances of female athletes, uncomfortable and objectifying uniforms, and appearance and competence-related teasing from male and female peers, as well as coaches.

To date, research has predominantly focused on athletes' perceptions of the extent to which coaches perpetuate athletes' body image concerns. However, several recent studies have been conducted exploring the perception of coaches and their role in addressing body image concerns among girls in sport. The findings of these studies indicate that although coaches are often able to identify body image concerns among their athletes, they are apprehensive to explicitly address these issues for fear of making the concerns worse. As such, systemic strategies are required within sport settings that upskill coaches as well as athletes and significant others in the athletes' environment to address body image concerns among adolescent girls in sport. At present, few such programs exist, and limited body image resources are available to coaches, despite coaches perceiving body image education as a personal and professional requirement for working with young people.

The current research will test the first online body image program for coaches. The Body Confident Coaching program was co-created with girls and coaches through an international multi-disciplinary partnership between academics, health professionals, industry, and community organizations. Multi-disciplinary partnerships can create a supportive landscape by upskilling athletes and coaches in dealing with body image concerns, which will likely lead to sustained sports participation and biopsychosocial benefits.

As such, the aim of the present study is to conduct a randomized controlled trial (RCT) to evaluate the effectiveness, feasibility, and acceptability of the Body Confident Coaching program. The program consists of five 20-minute modules that coaches complete online. Each session tackles a distinct theme related to body image in the sporting context. Outcomes will be assessed at pre- and post-intervention and include coaches' self-efficacy to tackle athletes' body image concerns (primary outcome), coaches' fat phobia and gender essentialist beliefs (secondary outcomes), and feasibility, acceptability, and adherence (process outcomes). The comparison control arm will be a waitlist control condition.

To undertake this project, coaches will be randomized into the intervention group or the control group, with 60 coaches anticipated in each arm. Those in the intervention condition will complete baseline assessments (target outcomes and demographic information), take part in the two-week intervention, and then complete the post-intervention assessments (target outcomes and feasibility and acceptability measures). Those in the waitlist control condition will complete the baseline assessments (target outcomes and demographic information) and a second assessment two weeks later (target outcomes only), after which they will get access to the online intervention. However, their engagement with the intervention will not be monitored or assessed. At completion of the post-intervention survey, all participants will receive a debrief form, outlining the study aims and objectives, and additional resources for body image and eating concerns. Lastly, to compensate participants for their time, coaches will receive an electronic voucher to the value of $25 dollars.

The investigators hypothesize that coaches who take part in the Body Confident Coaching intervention will report greater self-efficacy in identifying and tackling body image concerns among their athletes, and lower levels of fat phobia and gender essentialism at post-intervention than coaches who do not take part in the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Current coaches of adolescent girls
* English speaking
* US resident

Exclusion Criteria:

* Participants under 18 years of age
* Coaches outside of the US
* Coaches who only coach adult women or men/boys

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Change in coaches' self-efficacy in body image (assessed via the Coaches' Self-Efficacy in Body Image Scale) | Baseline, pre-intervention; immediately after the intervention (2 weeks later)
  The Coaches' Self-Efficacy in Body Image Scale (CSEBIS) assesses coaches' ability to describe, recognize, support, and prevent body image concerns among their athletes. CSEBIS scores range from 0-10 with higher scores on the CSEBIS indicating higher levels of self-efficacy.

SECONDARY OUTCOMES:
Change in coaches' fat phobia (assessed via the Fat Phobia Scale) | Baseline, pre-intervention; immediately after the intervention (2 weeks later)
  The Fat Phobia Scale (FPS) is a 14-item questionnaire regarding beliefs and feelings towards people who are fat or obese. FPS scores range from 1-5 with higher scores on the FPS indicating higher levels of fat phobia.
Change in coaches' gender essentialism (assessed via the Gender Essentialism Scale) | Baseline, pre-intervention; immediately after the intervention (2 weeks later)
  The Gender Essentialism Scale (GES) is a 25-item scale, rated from 1 (strongly disagree) to 5 (strongly agree), and assesses sex-role egalitarianism, support for discriminatory practices, and perceived fairness of gender-based treatment. GES scores range from 1-5 with higher scores on the GES indicating higher levels of gender essentialism.

OTHER OUTCOMES:
Total acceptability of the intervention (assessed via a self-report questionnaire) | Immediately after the intervention
  Coaches will complete feasibility and acceptability measures via a self-report questionnaire on a scale from 1 (Strongly Disagree) to 5 (Strongly Agree) within the following domains: 1) affective attitude (e.g., I liked this program); 2) burden (e.g., it was easy to follow the content of the program); 3) ethicality (e.g., I think this program is appropriate for coaches in my sport); 4) self-efficacy (e.g., I am confident that I will use the techniques I learned from this program); 5) perceived effectiveness (e.g., the program was successful in improving my knowledge about body image); and 6) content (e.g., how easy or difficult was it to follow the program?).
Total intervention adherence (assessed through session completion) | Immediately after the intervention
  Total intervention adherence will be assessed by the investigators as number of participants who complete the full intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Appearance Research, University of the West of England, Bristol, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guthold R, Stevens GA, Riley LM, Bull FC. Global trends in insufficient physical activity among adolescents: a pooled analysis of 298 population-based surveys with 1.6 million participants. Lancet Child Adolesc Health. 2020 Jan;4(1):23-35. doi: 10.1016/S2352-4642(19)30323-2. Epub 2019 Nov 21. PMID 31761562
- [Background] Koulanova, A., Sabiston, C. M., Pila, E., Brunet, J., Sylvester, B., Sandmeyer-Graves, A., & Maginn, D. (2021). Ideas for action: Exploring strategies to address body image concerns for adolescent girls involved in sport. Psychology of Sport and Exercise, 56, 102017.
- [Background] Neumark-Sztainer D, MacLehose RF, Watts AW, Pacanowski CR, Eisenberg ME. Yoga and body image: Findings from a large population-based study of young adults. Body Image. 2018 Mar;24:69-75. doi: 10.1016/j.bodyim.2017.12.003. Epub 2017 Dec 27. PMID 29288970
- [Background] Sabiston, C., Pila, E., Vani, M., & Thogersen-Ntoumani, C. (2019). Body image, physical activity, and sport: A scoping review. Psychology Of Sport And Exercise, 42, 48-57. doi: 10.1016/j.psychsport.2018.12.010
- [Background] Sabiston CM, Pila E, Crocker PRE, Mack DE, Wilson PM, Brunet J, Kowalski KC. Changes in body-related self-conscious emotions over time among youth female athletes. Body Image. 2020 Mar;32:24-33. doi: 10.1016/j.bodyim.2019.11.001. Epub 2019 Nov 14. PMID 31734408
- [Background] Slater A, Tiggemann M. Gender differences in adolescent sport participation, teasing, self-objectification and body image concerns. J Adolesc. 2011 Jun;34(3):455-63. doi: 10.1016/j.adolescence.2010.06.007. Epub 2010 Jul 31. PMID 20643477
- [Background] Vani MF, Pila E, Willson E, Sabiston CM. Body-related embarrassment: The overlooked self-conscious emotion. Body Image. 2020 Mar;32:14-23. doi: 10.1016/j.bodyim.2019.10.007. Epub 2019 Nov 13. PMID 31733410
- [Result] Schneider, J., Matheson, E. L., Tinoco, A., Gentili, C., White, P., Boucher, C., Silva-Breen, H., Goorevich, A., Diedrichs, P.C., & LaVoi, N. M. (2023). Body Confident Coaching: A pilot randomized controlled trial evaluating the acceptability of a web-based body image intervention for coaches of adolescent girls. Journal of Applied Sport Psychology. https://doi.org/10.1080/10413200.2023.2212023